CLINICAL TRIAL: NCT00820911
Title: An Extension to a 12-month, Open-label, Randomised, Multicenter, Sequential Cohort, Dose Finding Study to Evaluate the Efficacy, Safety and Tolerability of Oral AEB071 Versus Cyclosporine in Combination With Everolimus, Basiliximab and Corticosteroids in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of AEB071 Versus Cyclosporine in de Novo Renal Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEB071A2206E1; 2008-000531-18 (EudraCT Number)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplant; AEB071
MeSH Terms: interventions — Cyclosporine; Everolimus; sotrastaurin

ARMS (3):
- cyclosporine (reduced exposure) / everolimus (Active Comparator)
  Interventions: Drug: cyclosporine (reduced exposure) / everolimus
- AEB071 300 mg b.i.d. / everolimus (Experimental)
  Interventions: Drug: AEB071 300 mg b.i.d. / everolimus
- AEB071 200 mg b.i.d. / everolimus (Experimental)
  Interventions: Drug: AEB071 200 mg b.i.d. / everolimus

INTERVENTIONS:
Drug: cyclosporine (reduced exposure) / everolimus — twice daily
  Arms: cyclosporine (reduced exposure) / everolimus
Drug: AEB071 300 mg b.i.d. / everolimus — twice daily
  Arms: AEB071 300 mg b.i.d. / everolimus
Drug: AEB071 200 mg b.i.d. / everolimus — twice daily
  Arms: AEB071 200 mg b.i.d. / everolimus

SUMMARY:
This study will assess safety and efficacy of AEB071 combined with everolimus in a CNI-free (calcineurin inhibitor) regimen in renal transplant recipients.

ELIGIBILITY:
Inclusion criteria:

* Patient has been maintained on study drug for 12 months in the core study

Exclusion criteria:

* Not applicable
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
renal function as measured by the glomerular filtration rate (GFR) using the modification of diet in renal disease (MDRD) formula | at months 15, 18, 21, 24, 30, 36, 42, 48, 54 and 60 months after transplantation

SECONDARY OUTCOMES:
efficacy failure, defined as a composite efficacy endpoint of treated biopsy proven acute rejection, graft loss, death or loss to follow-up | at months 15, 18, 21, 24, 30, 36, 42, 48, 54 and 60 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Argentina (2):
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Clayton, Victoria
- Novartis Investigative Site, Innsbruck, Austria
- Novartis Investigative Site, Ghent, Belgium
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
- Novartis Investigative Site, Prague, Czechia
- France (3):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica, Slovakia
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Zurich, Switzerland, Switzerland
- Novartis Investigative Site, Taipei, Taiwan, Taiwan